CLINICAL TRIAL: NCT06342700
Title: A Randomized, Open-label, Single-dose, 4-period, 4--sequence, Crossover Phase I Relative Bioavailability Study Comparing Crystalline Formulation Tablet Versus Reference Amorphous Formulation Tablet of Rilzabrutinib (SAR444671) in Fasted and Fed Conditions in Healthy Male and Female Participants
Brief Title: A Food Effect and Relative Bioavailability Study of Rilzabrutinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PKM18138; U1111-1299-1906 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-03-18; First posted 2024-04-02 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Disorder; Healthy Volunteers
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: SAR444671 amorphous fasted (Active Comparator): Participants will receive single oral dose of amorphous tablet formulation rilzabrutinib (SAR444671) under fasted conditions on Day 1 for one period
  Interventions: Drug: Rilzabrutinib amorphous form
- Treatment B: SAR444671 crystalline fasted (Experimental): Participants will receive single oral dose of crystalline tablet formulation rilzabrutinib (SAR444671) under fasted conditions on Day 1 for one period
  Interventions: Drug: Rilzabrutinib crystalline form
- Treatment C: SAR444671 amorphous fed (Active Comparator): Participants will receive single oral dose of amorphous tablet formulation rilzabrutinib (SAR444671) under fed conditions on Day 1 for one period
  Interventions: Drug: Rilzabrutinib amorphous form
- Treatment D: SAR444671 crystalline fed (Experimental): Participants will receive single oral dose of crystalline tablet formulation rilzabrutinib (SAR444671) under fed conditions on Day 1 for one period
  Interventions: Drug: Rilzabrutinib crystalline form

INTERVENTIONS:
Drug: Rilzabrutinib crystalline form — Pharmaceutical form:Film coated tablet Route of administration:Oral
  Other Names: SAR444671
  Arms: Treatment B: SAR444671 crystalline fasted; Treatment D: SAR444671 crystalline fed
Drug: Rilzabrutinib amorphous form — Pharmaceutical form:Film coated tablet Route of administration:Oral
  Other Names: SAR444671
  Arms: Treatment A: SAR444671 amorphous fasted; Treatment C: SAR444671 amorphous fed

SUMMARY:
This is a cross-over, Phase 1, 4-arm study. The purpose of this study is to measure the relative bioavailability and food effect of crystalline formulation rilzabrutinib and amorphous formulation rilzabrutinib in healthy male and female participants aged 18 to 55 years of age.

The total study duration per participant is expected to be up to 36 days, including:

* Screening: up to 4 weeks
* Treatment periods: once successfully screened, enrolled participants will be randomized to 1 of 4 treatment sequences with 4 single dose treatment periods.
* Washout: One day washout is planned after each treatment period hence providing 2 days between doses.
* Safety follow-up: participants will be asked to participate in an end-of-study safety assessment upon discharge from the clinical study unit, ie, on Day 8 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50.0 and 100.0 kg, inclusive, if male, and between 40.0 and 90.0 kg, inclusive, if female, body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy participant. Hepatic transaminases (aspartate aminotransferase, alanine aminotransferase) should not exceed 1.25 × the upper laboratory norm (ULN); total bilirubin should not exceed 1 × ULN
* Willing to abstain from using tobacco or nicotine-containing products or consuming alcohol from check-in (Day -1) until discharge at end-of-study visit
* Willing to abstain from taking any prescription drugs, dietary supplements, or non-prescription drugs within 14 days or 5 half-lives, whichever, is longer, prior to the first dose of study drug through the follow-up phone call. Use of hormonal contraception and aspirin (at doses of ≤2000 mg/day) or ibuprofen (at doses of ≤1200 mg/day) are allowed prior to and during the study
* Negative urine drug/alcohol testing at screening and check-in (Day -1). Screening urine drug/alcohol testing may be repeated once if deemed appropriate by the site Investigator
* Willing to abstain from consuming grapefruit, star fruit, or Seville orange-containing products from 14 days prior to first dose of study drug until discharge from the clinical study unit

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynecologic (if female), infectious disease, or signs of acute illness
* Participant has clinical signs and symptoms consistent with COVID-19, eg, fever, dry cough, dyspnea, loss of taste and smell, sore throat, fatigue or confirmed infection by appropriate laboratory test within the last 4 weeks prior to Screening. Participant who had severe course of COVID-19 (ie, hospitalization, extracorporeal membrane oxygenation [ECMO], mechanically ventilated)
* Participant has a positive test result for SARS-CoV-2 (measured via Real-time Reverse Transcriptase Polymerase Chain Reaction [RT-PCR] or Rapid Antigen Test [RAT])
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month)
* Blood donation, any volume, within 1 month before inclusion
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure <30 mmHg within 3 minutes when changing from supine to standing position
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician. Participants with known hypersensitivity to any component of the IMP formulation or allergic disease diagnosed and treated by a physician
* History or presence of drug or alcohol abuse (alcohol consumption more than 40 g per day on a regular basis)
* Regular intake of nicotine (via patch, smoking, vaping or other forms) more than 10 mg per day (based on the average nicotine content of 10-12 mg of nicotine per cigarette and inhalation of up to 2 mg of nicotine per cigarette), and unable to stop smoking during the study (occasional smoker can be enrolled)
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day)
* If female, pregnancy (defined as positive β-HCG blood test), or breast-feeding
* Any medication (including St John's Wort or ginseng) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of aspirin/ibuprofen, hormonal contraception, and menopausal hormone replacement therapy
* Any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion:

  * Non-live vaccines, including COVID-19: last administration of a vaccine within 4 weeks before randomization
  * Live vaccines: last administration of a vaccine within 3 months before randomization
* Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab)
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates)
* Positive alcohol breath or alcohol urine test
* Positive pregnancy test
* Gilbert's Syndrome

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability as assessed by rilzabrutinib Cmax following administration of the test and reference formulations in the fasted state | Day 1 to Day 8
  Cmax: maximum plasma concentration
Relative bioavailability as assessed by rilzabrutinib AUClast following administration of the test and reference formulations in the fasted state | Day 1 to Day 8
  AUClast: area under the plasma concentration versus time curve from time zero to the last measurable concentration
Relative bioavailability as assessed by rilzabrutinib AUC following administration of the test and reference formulations in the fasted state | Day 1 to Day 8
  AUC: area under the plasma concentration versus time curve extrapolated to infinity

SECONDARY OUTCOMES:
Relative bioavailability as assessed by rilzabrutinib Cmax following administration of the test and reference formulations in the fed state | Day 1 to Day 8
  Cmax: maximum plasma concentration
Relative bioavailability as assessed by rilzabrutinib AUClast following administration of the test and reference formulations in the fed state | Day 1 to Day 8
  AUClast: area under the plasma concentration versus time curve from time zero to the last measurable concentration
Relative bioavailability as assessed by rilzabrutinib AUC following administration of the test and reference formulations in the fed state | Day 1 to Day 8
  AUC: area under the plasma concentration versus time curve extrapolated to infinity
Food effects as assessed by rilzabrutinib Cmax following administration of the test and reference formulations under the fed versus fasted state | Day 1 to Day 8
  Cmax: maximum plasma concentration
Food effects as assessed by rilzabrutinib AUClast following administration of the test and reference formulations under the fed versus fasted state | Day 1 to Day 8
  AUClast: area under the plasma concentration versus time curve from time zero to the last measurable concentration
Food effects as assessed by rilzabrutinib AUC following administration of the test and reference formulations under the fed versus fasted state | Day 1 to Day 8
  AUC: area under the plasma concentration versus time curve extrapolated to infinity
Number of participants with adverse events, treatment-emergent adverse events, serious adverse events and adverse events of special interest | Day 1 to Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Site Number : 8400001, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: PKM18138 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25706&tenant=MT_SNY_9011